CLINICAL TRIAL: NCT01704937
Title: Fecal Microbiota Transplant (FMT) for Relapsing C. Difficile Infection in Adults and Children Using a Frozen Inoculum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-P-001657
Record Dates: First submitted 2012-10-04; First posted 2012-10-12 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Clostridium Difficile Infection
Keywords: Fecal Microbiota Transplant; Clostridium difficile; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colonoscopy (Experimental): Fecal microbiota transplant ("stool transplant") from healthy, unrelated donor via colonoscopy
  Interventions: Drug: Fecal Microbiota Transplant (FMT)
- Nasogastric Tube (NGT) (Experimental): Fecal microbiota transplant ("stool transplant") from healthy, unrelated donor via NGT
  Interventions: Drug: Fecal Microbiota Transplant (FMT)

INTERVENTIONS:
Drug: Fecal Microbiota Transplant (FMT) — Reconstitution of normal flora by a "stool transplant" from a healthy individual to a C. difficile - infected recipient via colonoscopy or nasogastric tube

SUMMARY:
Fecal microbiota transplantation (FMT) is the reconstitution of normal flora by a "stool transplant" from a healthy individual to a C. difficile-infected recipient, and has long been a successful approach to recurrent/refractory C. difficile. The purpose of this project is to generate a frozen FMT inoculum from well-screened healthy volunteer donors which can be used repeatedly, particularly in those who do not have a healthy intimate partner or other related donor. Delivery of FMT has been performed colonoscopically, by fecal retention enema, or by the nasogastric route. This study will evaluate the safety and secondarily the efficacy of a frozen inoculum administered by nasogastric tube vs administered by colonoscope.

Subjects with recurrent/relapsing C. difficile infection (10 per group) will receive FMT via either:

* colonoscopy
* NGT

The primary endpoint is assessment of safety as measured by clinical events (GI, procedural, systemic). Efficacy will be defined as a resolution of diarrhea off antibiotics for C. difficile, in the absence of a need for OTHER systemic antibiotics, i.e. resumption of a normal bowel status for the individual. Secondary efficacy endpoints include weight, subjective well-being and relative clinical improvement per standardized questionnaire, and subject qualitative assessment of, and satisfaction with, the transplant procedures. Subjects will be monitored for clinical safety by history and standard exams and the follow-up questionnaire as well as followed closely by phone and in person.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or relapsing CDI defined as EITHER(13):

  * At least three episodes of mild-to-moderate CDI and failure of a 6-8 week taper with vancomycin with or without an alternative antibiotic (e.g. rifaximin, nitazoxanide).
  * At least two episodes of severe CDI resulting in hospitalization and associated with significant morbidity.
* Willingness to accept risk of unrelated donor stool
* Willingness to be randomized to NGT vs. colonoscopic delivery.
* Able to consent for self, or parental assent/child assent as age appropriate.

Exclusion Criteria:

* Anatomic contraindication to NGT
* Delayed gastric emptying syndrome
* Known chronic aspiration
* Contraindication to colonoscopy (ASA 4 or more)
* High risk of bacterial translocation (Immunosuppression, cirrhosis etc)
* Pregnant or breastfeeding women
* Acute unrelated infection or comorbid illness exaccerbation

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety | up to 6 mo post FMT
  Safety is assessed by clinical symptoms, exam, signs (GI and systemic)

SECONDARY OUTCOMES:
Efficacy | 3 months
  Efficacy is defined as resolution of C. Difficile signs and symptoms off antibiotics for C. difficile

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Hohmann, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Youngster I, Sauk J, Pindar C, Wilson RG, Kaplan JL, Smith MB, Alm EJ, Gevers D, Russell GH, Hohmann EL. Fecal microbiota transplant for relapsing Clostridium difficile infection using a frozen inoculum from unrelated donors: a randomized, open-label, controlled pilot study. Clin Infect Dis. 2014 Jun;58(11):1515-22. doi: 10.1093/cid/ciu135. Epub 2014 Apr 23. PMID 24762631